CLINICAL TRIAL: NCT02889991
Title: Comparative Study, Between Dry Needling Techniques, in the Evolution of Myofascial Pain Shoulder in Athletes. Elastography as Indicator in the Repair of Myofascial Tissue, Post-dry Needling.
Brief Title: Evolution of Myofascial Pain, Post-dry Needling. Repair and Measuring With Elastography, of Myofascial Tissue.
Acronym: INA-DMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Collaborators: FisioAraba Centre Physiotherapy S.C. (Unknown); Toshiba Medical Systems, S.A. (Unknown); Metron Medical Supplies S.L. (Unknown); Novasan, Medical & Health Products (Unknown)
Responsible Party: Principal Investigator, Francisco jiménez Hidalgo, Physiotherapist, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: M10_2015_142_GRANADOS
Record Dates: First submitted 2016-07-26; First posted 2016-09-07 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2017-08

CONDITIONS: Myofascial Pain Syndromes; Dry Needling, Technique for the Treatment of the Myofascial Trigger Points; Elastography
Keywords: Myofascial pain.; Myofascial trigger point.; Infraspinatus muscle.; Deep dry needling.; Local twitch response.; Fascial mechanotransduction.; Needle grasp.; Myofascial fibrosis.; Elastography.
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High Intensity Dry Needling (Experimental): Maneuver of Input-Output with the acupuncture needle, until the disappearance of local twitch responses or patient tolerance.
  Interventions: Other: High Intensity Dry Needling
- Low Intensity Dry Needling (Experimental): Maximum 10 input-output maneuvers with acupuncture needle or maximum 3 local twitch responses or patient tolerance.
  Interventions: Other: Low intensity Dry Needling
- Fascial mechanotransduction Dry needling (Experimental): Maneuver of input, screwing and pulling out of the needle acupuncture.
  Interventions: Other: Fascial Mechanotransduction Dry Needling
- Placebo Dry Needling Technique (Sham Comparator): Technique is performed with the "Park´s Sham device".
  Interventions: Other: Technique Placebo of Dry Needling

INTERVENTIONS:
Other: High Intensity Dry Needling — This technique follows the criteria established by Dr Hong C-Z. This technique is known as "fast in and fast out technique" and uses repeated insertion of the acupuncture needle in the myofascial trigger point, with the aim to get multiple local twitch responses. The technique ends when the local twitch responses disappear.
  Arms: High Intensity Dry Needling
Other: Low intensity Dry Needling — Technique proposed by the main investigator and based on the studies of Professor Dr. Jay P. Shah and the mechanisms of neuromodulation that transmits us the acupuncture scientific evidence.
  Arms: Low Intensity Dry Needling
Other: Fascial Mechanotransduction Dry Needling — The Fascial Mechanotransduction Dry Needling Technique, strikes with the acupuncture needle until it reaches and pierces the myofascial trigger point. Then the acupuncture needle is rolled in the connective tissue, which causes an intense coupler that we define as "needle grasp". Finally, the acupuncture needling is pulled-out twice.
  The screwing and the two pull-out of the acupuncture needle is performed in the infraspinatus and supraspinatus muscles and we describe it as mechanotransduction cycle. Each cycle lasts 30 seconds and the whole technique lasts 3 minutes per session.
  Arms: Fascial mechanotransduction Dry needling
Other: Technique Placebo of Dry Needling — Technique with a total duration of 3 minutes per session:
  * To locate the myofascial trigger points of infraspinatus and supraspinatus muscles and put each bridle on them.
  * Monitor longitudinally taut band, with index and middle fingers.
  * Percuss with tube and needle placebo (Sham needle) on Infraspinatus.
  * Remove the tube and needle placebo from the device. Reintroducing the placebo needle into the tube and strike on the supraspinatus. Repeat this sequence without interruption for 3 minutes.
  * Remove the bridles and perform hemostasis with cotton.
  * We will give end to the technique placebo of dry needling.
  Other Names: Control Group
  Arms: Placebo Dry Needling Technique

SUMMARY:
This study evaluates the deep dry needling technique as a percutaneous technique included in the professional field of physiotherapy.

The project quantifies a significant limit on the number of local twitch responses necessary for the favorable treatment of myofascial pain and analyzes the injury degree and/or the repair of myofascial tissue, with "Elastography".

DETAILED DESCRIPTION:
The myofascial shoulder pain caused by myofascial trigger points, is one of the main causes of medical consultation and functional disability in the general population and particularly in the amateur athlete.

Nowadays, many physiotherapists all over the world, study and practice the dry needling as a therapeutic tool for the treatment of myofascial trigger points. The most used modality is the technique described by Hong:

* This technique introduces an acupuncture needle in the skin until reaching the dysfunctional muscle fiber. To do so, it uses maneuvers "fast in" and "fast out" of needle, until the extinction of local twitch responses or the tolerance of the patient.
* The local twitch response is defined as a reflex and transitory contraction of a group of muscle fibers associated with a myofascial trigger points.
* The technique eliminates muscle contractile activity by mechanical interruption of their muscle fibers, mechanism which finishes with the sensitization of nearby nerves and with the start of the nociceptive modulation peripheral, segmental and central.

The dry needling technique, in its eagerness to obtain local twitch responses, pierces the muscle fibers both dysfunctional and normal, the fascial tissue that wraps the myofascial trigger points and also neuro-vascular structures. That is, the treatment of myofascial trigger points with dry needling, makes reference to a mechanical trauma done with a acupuncture needle.

The myofascial tissue injured can suffer repair or regeneration, which is mainly due to the extension of the lesion. The process of healing of a wound is strictly regulated by multiple growth factors and cytokines, which are released into the wound. The alterations that disturb the healing process, can lead to chronic wounds that do not heal or to an excessive fibrosis.

The pathobiological processes, in form of fibrosis, would present changes in stiffness and elasticity of the neo-tissue. The quantitative elastography, is shown as an effective tool to measure the amount of fibrosis, occasioned by repeated percussion of the acupuncture needle on the myofascial tissue.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral shoulder pain or referred pain pattern of the infraspinatus muscle.
* Pain Intensity with a minimum score of 2 on the Wong-Baker scale, using the homolateral "test hand-back".
* Process time more than 1 and less than 10 weeks.
* Age of 18 years old to 49 years old.
* Written Informed Form.

Exclusion Criteria:

* Conventional pharmacological treatment of NSAIDs and / or muscle relaxants, the 48 hours before or during the study.
* Coagulation pathology or anticoagulant therapy.
* Pretreatment with infiltration and / or steroid injections during the last year.
* Physiotherapy Pretreatment, in the cervical region or shoulder girdle during or in the last week taking part in the study.
* Dry needling pretreatment in the cervical region and / or shoulder girdle during or in the last month before taking part in the study.
* History of fracture or dislocation of the shoulder to study, in the last year.
* Dermatological disorders or erosions in the treatment area (infraspinatus fossa).
* Metals allergy such as chromium or nickel.
* Fibromyalgia diagnosis, myelopathy, cervical radiculopathy or neurologic disease.
* Fear of needles.
* Pregnant women.
* Suffering a traumatic accident of the upper extremity and / or cervical-thoracic spine during the study (it will pass to the zero week).
* Medical-legal litigious, by financial compensation.
* Drugs or alcohol abuse / consumption history.
* Cognitive inability to complete the health forms.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2017-01-28 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Number of input-output of acupuncture needle in the infraspinatus and supraspinatus muscles. | Three interventions during 40 days.
  This outcome only used with High Intensity Dry Needling and Low Intensity Dry Needling techniques.
  The number of input-output of the acupuncture needle are established in each technique.
  The first 3 interventions are recorded with a compact sporty camera with a bracket on the head. This method allows recording, specifically, the number of input-output of the acupuncture needle.
Number of local twitch response in the infraspinatus and supraspinatus muscles. | Three interventions during 40 days.
  The limits of number of local twitch response are established in each technique to study.

SECONDARY OUTCOMES:
Active joint range of motion | Four interventions during 40 days.
  This dependent variable is measured before and after each intervention. We assign the following reference: Active joint range of motion - flexion, Active joint range of motion - abduction, Active joint range of motion - internal rotation and Active joint range of motion - external rotation.
Feeling of shoulder pain | Four interventions during 40 days.
  This dependent variable is measured before and after each intervention. We used the "hand-back test" and measure the pain feeling with the Wong-Baker scale. Score 0-5 (0 = No pain, 5 = Hurts worst)
Life quality related to health shoulder. | Two interventions during 40 days.
  We measure the shoulder disability in the daily life activities, at work and practising sports with the questionnaire "Disabilities of the Arm, Shoulder and Hand (DASH)"
Pressure pain threshold | Four interventions during 40 days.
  This dependent variable is measured before and after each intervention. We use the electronic algometer as a measurement tool.
Quality of the myofascial tissue by elastography | Two interventions during 40 days. A third intervention at 6 months after the second, to determine the degree of myofascial fibrosis.
  Check with quantitative elastography, the presence or not of fibrosis and / or repair of the myofascial tissue.

OTHER OUTCOMES:
Laterality | One intervention during 40 days.
  Indicate which is the injured shoulder (Left or right)
Age | One intervention during 40 days.
  Indicate patient´s years old
Sex | One intervention during 40 days.
  Indicate patient´s sex (Male/Female)
Chronicity of pain | One intervention during 40 days.
  Indicate how long the patient suffers shoulder pain.
Presence of referred pain pattern in the infraspinatus muscle | Two interventions during 40 days.
  Indicate the presence of referred pain pattern (Yes or No)
Myofascial trigger points related to shoulder pain | Two interventions during 40 days.
  Indicate which are the muscles related to shoulder pain.
Practice sport? | One intervention during 40 days.
  Indicate if patient practices sport (Yes or No)
Sport discipline | One intervention during 40 days.
  Indicate which sport discipline practices the patient.
Sporty feature | One intervention during 40 days.
  Indicate if the patient uses the shoulder in the sport (Yes or No).
Years of sport practice | One intervention during 40 days.
  Indicate the number of years practising the sport.
Hours per week | One intervention during 40 days.
  Indicate how many hours per week does the patient practises the sport.
Professional activity | One intervention during 40 days.
  Indicate if the patient lifts up or not the upper limb, over 90 ° of flexion and / or abduction in his or her job (Yes or No).
Accident during the treatment | One intervention during 40 days.
  Indicate if the patient has suffer any accident during the treatment (Yes or No)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Jiménez, PT, Principal Investigator — University of Basque Country
Locations (1):
- Physiotherapy Centre FISIOARABA, Vitoria-Gasteiz, Alava, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Page P. Shoulder muscle imbalance and subacromial impingement syndrome in overhead athletes. Int J Sports Phys Ther. 2011 Mar;6(1):51-8. PMID 21655457
- [Background] Hong CZ. New trends in myofascial pain syndrome. Zhonghua Yi Xue Za Zhi (Taipei). 2002 Nov;65(11):501-12. PMID 12583512
- [Background] Hong CZ. Lidocaine injection versus dry needling to myofascial trigger point. The importance of the local twitch response. Am J Phys Med Rehabil. 1994 Jul-Aug;73(4):256-63. doi: 10.1097/00002060-199407000-00006. PMID 8043247
- [Background] Gerwin RD, Dommerholt J, Shah JP. An expansion of Simons' integrated hypothesis of trigger point formation. Curr Pain Headache Rep. 2004 Dec;8(6):468-75. doi: 10.1007/s11916-004-0069-x. PMID 15509461
- [Background] Cotchett MP, Landorf KB, Munteanu SE. Effectiveness of dry needling and injections of myofascial trigger points associated with plantar heel pain: a systematic review. J Foot Ankle Res. 2010 Sep 1;3:18. doi: 10.1186/1757-1146-3-18. PMID 20807448
- [Background] Huang YT, Lin SY, Neoh CA, Wang KY, Jean YH, Shi HY. Dry needling for myofascial pain: prognostic factors. J Altern Complement Med. 2011 Aug;17(8):755-62. doi: 10.1089/acm.2010.0374. Epub 2011 Jul 11. PMID 21745098
- [Background] Ay S, Evcik D, Tur BS. Comparison of injection methods in myofascial pain syndrome: a randomized controlled trial. Clin Rheumatol. 2010 Jan;29(1):19-23. doi: 10.1007/s10067-009-1307-8. Epub 2009 Oct 20. PMID 19838864
- [Background] Tough EA, White AR, Cummings TM, Richards SH, Campbell JL. Acupuncture and dry needling in the management of myofascial trigger point pain: a systematic review and meta-analysis of randomised controlled trials. Eur J Pain. 2009 Jan;13(1):3-10. doi: 10.1016/j.ejpain.2008.02.006. Epub 2008 Apr 18. PMID 18395479
- [Background] Hsieh YL, Yang SA, Yang CC, Chou LW. Dry needling at myofascial trigger spots of rabbit skeletal muscles modulates the biochemicals associated with pain, inflammation, and hypoxia. Evid Based Complement Alternat Med. 2012;2012:342165. doi: 10.1155/2012/342165. Epub 2012 Dec 23. PMID 23346198
- [Background] Tekin L, Akarsu S, Durmus O, Cakar E, Dincer U, Kiralp MZ. The effect of dry needling in the treatment of myofascial pain syndrome: a randomized double-blinded placebo-controlled trial. Clin Rheumatol. 2013 Mar;32(3):309-15. doi: 10.1007/s10067-012-2112-3. Epub 2012 Nov 9. PMID 23138883
- [Background] Midwood KS, Williams LV, Schwarzbauer JE. Tissue repair and the dynamics of the extracellular matrix. Int J Biochem Cell Biol. 2004 Jun;36(6):1031-7. doi: 10.1016/j.biocel.2003.12.003. PMID 15094118
- [Background] Jarvinen TA, Jarvinen TL, Kaariainen M, Kalimo H, Jarvinen M. Muscle injuries: biology and treatment. Am J Sports Med. 2005 May;33(5):745-64. doi: 10.1177/0363546505274714. PMID 15851777
- [Background] Domingo A, Mayoral O, Monterde S, Santafe MM. Neuromuscular damage and repair after dry needling in mice. Evid Based Complement Alternat Med. 2013;2013:260806. doi: 10.1155/2013/260806. Epub 2013 Apr 9. PMID 23662122
- [Background] Sikdar S, Shah JP, Gebreab T, Yen RH, Gilliams E, Danoff J, Gerber LH. Novel applications of ultrasound technology to visualize and characterize myofascial trigger points and surrounding soft tissue. Arch Phys Med Rehabil. 2009 Nov;90(11):1829-38. doi: 10.1016/j.apmr.2009.04.015. PMID 19887205
- [Background] Langevin HM, Nedergaard M, Howe AK. Cellular control of connective tissue matrix tension. J Cell Biochem. 2013 Aug;114(8):1714-9. doi: 10.1002/jcb.24521. PMID 23444198
- [Background] Ingber DE, Wang N, Stamenovic D. Tensegrity, cellular biophysics, and the mechanics of living systems. Rep Prog Phys. 2014 Apr;77(4):046603. doi: 10.1088/0034-4885/77/4/046603. PMID 24695087
- [Background] Shah JP, Gilliams EA. Uncovering the biochemical milieu of myofascial trigger points using in vivo microdialysis: an application of muscle pain concepts to myofascial pain syndrome. J Bodyw Mov Ther. 2008 Oct;12(4):371-384. doi: 10.1016/j.jbmt.2008.06.006. Epub 2008 Aug 13. PMID 19083696
- [Background] Leung L. Neurophysiological basis of acupuncture-induced analgesia--an updated review. J Acupunct Meridian Stud. 2012 Dec;5(6):261-70. doi: 10.1016/j.jams.2012.07.017. Epub 2012 Aug 22. PMID 23265077